CLINICAL TRIAL: NCT00413153
Title: Metabolic Effects of Switching Kaletra to Boosted Reyataz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Steven K. Grinspoon, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-P-002239
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV; Kaletra; Reyataz; Insulin sensitivity; Lipids; Body Composition; Receiving Kaletra; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Insulin Resistance | interventions — atazanavir, ritonavir drug combination; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Boosted Reyataz (300mg atazanavir + 100mg ritonavir)
  Interventions: Drug: atazanavir/ritonavir
- 2 (Active Comparator): Kaletra (pre-study dose)
  Interventions: Drug: lopinavir/ritonavir

INTERVENTIONS:
Drug: atazanavir/ritonavir — atazanavir 300mg + ritonavir 100mg once daily
  Other Names: Boosted Reyataz
  Arms: 1
Drug: lopinavir/ritonavir — patient remains on their pre-study dose of lopinavir/ritonavir
  Other Names: Kaletra
  Arms: 2

SUMMARY:
To study the effects of switching from Kaletra to Boosted Reyataz on glucose, lipids and fat in HIV-infected patients.

DETAILED DESCRIPTION:
The primary objective of this study is to determine tissue specific glucose trafficking in patients before and after switching from a regimen containing Lopinavir/ritonavir (LPV/r) to one containing atazanavir/ritonavir (ATV/r). Secondary outcome measures of interest will include insulin sensitivity determined by clamp testing, and lipid metabolism and hepatic glucose production assessed using stable isotope techniques. We hypothesize that switching protease inhibitor (PI) to ATV/r from LPV/r will result in direct increases in glucose uptake in muscle and visceral adipose tissue in association with improvements in overall whole body insulin sensitivity compared to remaining on LPV/r. We will complete a prospective randomized trial of Human Immunodeficiency Virus (HIV) infected patients who have been on a stable antiretroviral (ARV) regimen containing LPV/r for at least 6 months and who will be randomized to either switch to a regimen containing ATV/r or remain on LPV/r for 6 months. Each subject will complete Positron Emission Tomography (PET) 18-fluorodeoxyglucose (FDG) imaging during a hyperinsulinemic clamp study at baseline and 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed HIV infection
2. Age between 18-65 years
3. Stable antiviral regimen containing at least 2 nucleoside reverse transcriptase inhibitors (NRTI's) and LPV/r for ³ 6 mos
4. CD4 count > 400 cell/mm3
5. Metabolic complication as indicated by one or more of hyperinsulinemia (fasting insulin >= 15 mIU/ml), hypercholesteremia (fasting total cholesterol >= 200 mg/dL), hypertriglyceridemia (fasting triglycerides >= 150 mg/dL), or treatment with a lipid lowering medication.

Exclusion Criteria:

1. Hemoglobin < 11.0 g/dL
2. History of Diabetes Mellitus
3. Currently on medication for Diabetes
4. Therapy with glucocorticoid, growth hormone or other anabolic agents currently or within the past 3 months
5. Current substance abuse, including alcohol, cocaine and/or heroin
6. Any contraindication to ATV/r or known allergy to ATV
7. Concurrent therapy with: Bepridil; cisapride; ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine); indinavir; irinotecan; lovastatin; midazolam; pimozide; proton pump inhibitors (esomeprazole, lansoprazole, omeprazole); rifampin; simvastatin; St John's wort; or triazolam
8. New or serious opportunistic infection in the past 3 months
9. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Stanley TL, Joy T, Hadigan CM, Liebau JG, Makimura H, Chen CY, Thomas BJ, Weise SB, Robbins GK, Grinspoon SK. Effects of switching from lopinavir/ritonavir to atazanavir/ritonavir on muscle glucose uptake and visceral fat in HIV-infected patients. AIDS. 2009 Jul 17;23(11):1349-57. doi: 10.1097/QAD.0b013e32832ba904. PMID 19474651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through information given to HIV-care providers, postings in HIV-community organizations, newspaper advertisements, and the Massachusetts General Hospital research patient data registry. Recruitment began in March, 2006, and continued through May, 2008.
Pre-assignment Details: After screening visit to determine eligibility, subjects were asked to continue their current antiretroviral medications until the baseline visit, immediately after which they were randomized to continue lopinavir/ritonavir or switch to atazanavir/ritonavir.
Groups:
- Boosted Reyataz (ATV/r): Boosted Reyataz (300mg atazanavir + 100mg ritonavir)
- Continue Kaletra (LPV/r): Kaletra (pre-study dose)
Period: Overall Study
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Started | 7 | 8
Completed | 5 | 7
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r) | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (8) | 50 (6) | 48 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Glucose Trafficking
Description: 6 month mean and standard deviation for glucose uptake into anterior thigh muscle as measured by FDG/PET scanning during euglycemic hyperinsulinemic clamp. During the hyperinsulinemic conditions of the clamp, glucose and 18-FDG [labeled glucose] are taken up by muscle. The quantity of 18-FDG taken up is measured by the PET scan. Although there are no well-accepted norms for this measurement, a higher value indicates that more glucose is being taken up by (or "trafficked to") muscle. Increased uptake of glucose indicates increased muscle insulin sensitivity.
Time Frame: 6 months
Population: Only data from subjects with 0 and 6 month Positron Emission Tomography (PET) scans were analyzed.
Measure: Mean (Standard Deviation); unit: umol/kg/min
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 6
umol/kg/min | 26.7 (8.1) | 24.4 (17.7)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); Initial samples size of N=16 calculated to provide 80% power to detect a 30% change in muscle glucose uptake between groups. Student's t-test used to compare change from baseline and determine treatment effect (net difference over time between the ATV/r vs. LPV/r groups); Test type: Superiority or Other; p = 0.035, t-test, 2 sided

2. Secondary Outcome: Insulin Sensitivity
Description: 6 month mean and standard deviation for insulin-stimulated glucose uptake (M) per unit insulin at 120 minutes as measured by euglycemic hyperinsulinemic clamp.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: umol/kg/min per uU/mL insulin
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
umol/kg/min per uU/mL insulin | 39.0 (17.7) | 49.2 (22.5)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); Repeated measures ANCOVA, controlling for baseline values, used to assess treatment effect of the randomization over 6 months (net difference over time between ATV/r vs. LPV/r); Test type: Superiority or Other; p = 0.12, Repeated measures ANCOVA

3. Secondary Outcome: Fasting Glucose
Description: 6 month mean and standard deviation for fasting glucose.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
mg/dL | 84 (7) | 90 (21)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); Repeated measures ANCOVA, controlling for baseline values, used to assess treatment effect of the randomization over 6 months (net difference over time between ATV/r vs.LPV/r); Test type: Superiority or Other; p = 0.002, Repeated Measures ANCOVA

4. Secondary Outcome: Lipid Metabolism - Serum Triglyceride
Description: 6 month mean and standard deviation for serum triglyceride.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
mg/dL | 147 (92) | 209 (87)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.02, Repeated measures ANCOVA

5. Secondary Outcome: Body Composition - Visceral Adipose Tissue
Description: 6 month mean and standard deviation for visceral adipose tissue (VAT) as measured by single slice computed tomography (CT) scan at the L4 pedicle (pedicle of 4th lumbar vertebra).
Time Frame: 6 months
Population: Data from participants with 0 & 6 month data analyzed.
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
square centimeters | 91 (34) | 167 (61)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); Test type: Superiority or Other; p = 0.047, t-test, 2 sided

6. Secondary Outcome: Immune Parameters -- CD4 Count
Description: 6 month mean and standard deviation for CD4+ count.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: cells/microL
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
cells/microL | 432 (192) | 688 (230)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.72, Repeated Measures ANCOVA

7. Secondary Outcome: Liver Enzymes -- Aspartate Aminotransferase (AST)
Description: 6 month mean and standard deviation for AST.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
U/L | 39 (29) | 42 (29)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.22, Repeated Measures ANCOVA

8. Secondary Outcome: Liver Enzymes -- Alanine Aminotransferase (ALT)
Description: 6 month mean and standard deviation for ALT.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
U/L | 61 (29) | 65 (34)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.004, Repeated Measures Ancova

9. Secondary Outcome: Total Bilirubin
Description: 6 month mean and standard deviation for total bilirubin.
Time Frame: 6 months
Population: Repeated measures analysis using all available data points for each participant
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Number analyzed (Participants) | 5 | 7
mg/dL | 2.8 (2.7) | 0.6 (0.3)
Statistical Analysis 1: Comparison: Boosted Reyataz (ATV/r) vs Continue Kaletra (LPV/r); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0002, Repeated Measures ANCOVA

ADVERSE EVENTS:
Time Frame: 6 month study period
Description: All subjects had physical examinations and were queried about any adverse event at each study visit (baseline, 2 weeks, 1 month, 2 months, 4 months, and 6 months), and bilirubin, ALT, ALT, CD4+ count, and HIV ultrasensitive viral load were sent at all of these timepoints.
Arm/Group | Boosted Reyataz (ATV/r) | Continue Kaletra (LPV/r)
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/8
Other Adverse Events (participants affected / at risk) | 6/7 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boosted Reyataz (ATV/r) (N=7) | Continue Kaletra (LPV/r) (N=8)
Giardia Lamblia Infection (Gastrointestinal disorders) | 1 (1) | 0 (0) — hospitalization required for Giardia lamblia infection
Mental Status Changes (General disorders) | 1 (1) | 0 (0) — Mental status changes requiring hospitalization, found to be caused by combination of prescribed opiates
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boosted Reyataz (ATV/r) (N=7) | Continue Kaletra (LPV/r) (N=8)
cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
hyperbilirubinemia (Gastrointestinal disorders) | 6 | 0
HIV RNA Copy Number Increased (Infections and infestations) | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0
transaminitis (Gastrointestinal disorders) | 1 | 0 — ALT and/or AST elevated to any degree above the upper limit of normal.
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less